CLINICAL TRIAL: NCT04652531
Title: Autologous Serum-derived Extracellular Vesicles to Treat Venous Trophic Lesions Not Responsive to Conventional Treatments
Brief Title: Autologous Serum-derived EV for Venous Trophic Lesions Not Responsive to Conventional Treatments
Acronym: SER-VES-HEAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Maria Felice Brizzi, Associate Professor, University of Turin, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS2/1095/0090491
Record Dates: First submitted 2020-11-23; First posted 2020-12-03 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Ulcer Venous
Keywords: Autologous EV; serum; ulcers; vascular disease
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Peri-wound injection of the vesicles will be performed in a sterile environment. Sterile gauze and an elastic-compression bandage will be applied. The contralateral ulcer will be treated with a standard dressing and an elastic compression bandage. The patients will be evaluated on an outpatient basis on day 3 and then weekly.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): In the treatment arm, the lesion will be treated with EV for 3 weeks once a week
  Interventions: Other: Autologous extracellular vesicles from serum
- Internal control (Sham Comparator): The contralateral ulcer will be treated with a standard dressing and an elastic-compression bandage for 3 weeks.
  Interventions: Other: Autologous extracellular vesicles from serum

INTERVENTIONS:
Other: Autologous extracellular vesicles from serum — Peri-wound injection of the vesicles will be performed in a sterile environment. Sterile gauze and an elastic-compression bandage will be applied.

SUMMARY:
Venous ulcers are defined by the presence of open lesions which represent the final stage of chronic venous disease or post-thrombotic syndrome. The risk factors for the development of venous ulcers include age, obesity, female sex, trauma, immobility, factor V mutation, thrombosis, venous agenesis.

Recommendation by the current guidelines includes compression and advanced dressing. However, in several cases, they fail to change patients' outcome. The aim of this study is to identify an alternative therapy to treat venous trophic lesions not responding to traditional therapeutic approaches using extracellular vesicles obtained from autologous serum.

DETAILED DESCRIPTION:
In recent years, several in vitro and in vivo studies have provided been the beneficial effects of stem cells for tissue regeneration. Moreover, several randomized trials are ongoing and the interim results seem to give promising results and indicate their safety. Alternative approaches have recently been proposed, such as the injection of platelet preparation or the use of acellular amniotic membranes or extracellular vesicles (EV). EV act as cell-to-cell paracrine or endocrine-like communication mechanisms. The therapeutic potential of EV depends on the transfer of their cargo(proteins, RNAs, DNA, lipids, etc) to target cells (1). In the last decades, several pre-clinical studies have demonstrated safety. A pilot study was recently published on the use of EV as an effective treatment for retinal damage. At the University of Turin using a mouse model of ischemia/ reperfusion of the lower limb it was demonstrated that the intramuscular administration of EV obtained from the serum of healthy donors was associated with a higher density of local capillaries and an increase in laser Doppler signal compared to controls (2). A simple in vitro functional potency assay was developed, which allowed predicting EV therapeutic efficacy in vivo. The best response was obtained by intravenous administration immediately after surgical ligation and intramuscular in the next two days (T1 and T2). Through the Laser Doppler study, distal perfusion was evaluated after 7 days, which showed a clear improvement and protection of muscle damage. A more recent study has shown that even subjects with high cardiovascular risk (diabetic, obese, diabetic/obese and with arterial disease of the lower limbs) can benefit from the use of autologous EV (3).

The pilot study will involve the enrollment of 10 patients with bilateral venous ulcer refractory to conventional treatment for more than 6 months, recruited at the Vascular Ulcer Clinic of University Vascular Surgery. At the time of recruitment, venous Eco Doppler will be performed to evaluate the superficial and deep venous and arterial system to exclude possible "mixed" etiologies. A blood sample will then recovered for EV isolation in collaboration with the Blood Bank of the City of Health and Science of Turin. The characteristics of the ulcer will be entered in the database: dimensions (photo), margins, bottom and a swab for microbiology will be performed. Patients whose swab will be positive will be excluded.

EV will be analysed for their biological activity using the potency assay and will be used only if found to be effective (potency test). Subsequently, peri-wound injection of EV will be performed in a sterile environment. Sterile gauze and an elastic-compression bandage will be applied. As an internal control, the contralateral ulcer will be treated with a standard dressing and an elastic compression bandage. The patients will be evaluated on an outpatient basis on day 3 and then weekly. The results of treated patients will be collected in a dedicated database.

ELIGIBILITY:
Inclusion Criteria: Adults and conscious patients

-

Exclusion Criteria:

* :> 85 years, diabetics, autoimmune diseases, neoplastic, arterial disease of the lower limbs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the ulcer area from baseline to eight weeks | 8 weeks
  Ulcer areas will be recorded at baseline and weekly using digital camera. A standard rule was positioned on the surface of the skin around the ulcers to standardize the images and to allow data analysis. The ImageJ analysis program will be used to calculate the ulcer area. A blinded investigator manually delimitated the ulcer area to calculate the area. The total area will be expressed in square centimeters.

SECONDARY OUTCOMES:
Pain change | 8 week
  All patients should record their subjective feelings, including pain, burning and secretions. The level of pain will be monitored during the treatment as patient's experienced pain (decrease, unchange and/or increase). The amount of secretion will be classified as follow: absent, small, moderate, or abundant.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Felice Brizzi, MD, Principal Investigator — University of Turin, Italy; Giovanni Camussi, MD, Study Chair — University of Turin, Italy
Locations (1):
- AOU San Giovanni Battista, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kholia S, Ranghino A, Garnieri P, Lopatina T, Deregibus MC, Rispoli P, Brizzi MF, Camussi G. Extracellular vesicles as new players in angiogenesis. Vascul Pharmacol. 2016 Nov;86:64-70. doi: 10.1016/j.vph.2016.03.005. Epub 2016 Mar 22. PMID 27013016
- [Result] Cavallari C, Ranghino A, Tapparo M, Cedrino M, Figliolini F, Grange C, Giannachi V, Garneri P, Deregibus MC, Collino F, Rispoli P, Camussi G, Brizzi MF. Serum-derived extracellular vesicles (EVs) impact on vascular remodeling and prevent muscle damage in acute hind limb ischemia. Sci Rep. 2017 Aug 15;7(1):8180. doi: 10.1038/s41598-017-08250-0. PMID 28811546
- [Result] Cavallari C, Figliolini F, Tapparo M, Cedrino M, Trevisan A, Positello L, Rispoli P, Solini A, Migliaretti G, Camussi G, Brizzi MF. miR-130a and Tgfbeta Content in Extracellular Vesicles Derived from the Serum of Subjects at High Cardiovascular Risk Predicts their In-Vivo Angiogenic Potential. Sci Rep. 2020 Jan 20;10(1):706. doi: 10.1038/s41598-019-55783-7. PMID 31959759